CLINICAL TRIAL: NCT01917617
Title: The Feasibility Study of Oral Rehydration Therapy for Short Hydration in Chemotherapy With Cisplatin Plus Gemcitabine for Biliary Tract Cancer
Brief Title: Oral Rehydration Therapy for Short Hydration in Chemotherapy With CDDP Plus GEM for Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHBO1302; UMIN000010695 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-08-04; First posted 2013-08-06 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2017-05

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; World Health Organization oral rehydration solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral rehydration group（Short Hydration） (Experimental): Gemcitabine； gemzer Cisplatin；Cispulan Oral Rehydration Solution(ORS)；OS-1
  Short hydration via oral rehydration solution (OS-1)
  Cisplatin plus gemcitabine will be administered via infusion as follows; 500 ml of 0.9% saline including cisplatin (25 mg per square meter of body-surface area) over 1 hour followed by 250 ml of 0.9% saline including gemcitabine over 30 minutes. Before and after the infusion, each 500ml bottle of oral rehydration solution (OS-1) will be taken respectively.
  Interventions: Drug: Gemcitabine , Cisplatin, Oral Rehydration Solution (ORS)
- Standard group（Long Hydration） (Active Comparator): Drug: Gemcitabine , Cisplatin
  Other Names:
  Gemcitabine； gemzer Cisplatin； Cispulan
  Standard hydration via intravenous infusion
  Cisplatin plus gemcitabine will be administered via usual infusion regimen by each hospital. In general, it is administered total 2 litters over 3 hours or more.
  Interventions: Drug: Gemcitabine , Cisplatin

INTERVENTIONS:
Drug: Gemcitabine , Cisplatin, Oral Rehydration Solution (ORS) — Short hydration via oral rehydration solution (OS-1)
  Cisplatin plus gemcitabine will be administered via infusion as follows; 500 ml of 0.9% saline including cisplatin (25 mg per square meter of body-surface area) over 1 hour followed by 250 ml of 0.9% saline including gemcitabine over 30 minutes. Before and after the infusion, each 500ml bottle of oral rehydration solution (OS-1) will be taken respectively.
  Other Names: Gemcitabine； gemzer; Cisplatin；Cispulan; Oral Rehydration Solution(ORS)；OS-1
  Arms: Oral rehydration group（Short Hydration）
Drug: Gemcitabine , Cisplatin — Standard hydration via intravenous infusion
  Cisplatin plus gemcitabine will be administered via usual infusion regimen by each hospital. In general, it is administered total 2 litters over 3 hours or more.
  Other Names: Gemcitabine； gemzer; Cisplatin； Cispulan
  Arms: Standard group（Long Hydration）

SUMMARY:
The objective of this study is to evaluate the safety and feasibility of oral rehydration therapy for short hydration in patients with biliary tract cancer who will undergo the chemotherapy including gemcitabine and cisplatin.

DETAILED DESCRIPTION:
A large amount of fluid infusion is required to load for the prevention of renal dysfunction by Cisplatin in combination of GC therapy. There is a problem infusion time is take a long time for this. In many institutions in Japan, GC therapy is performed over 3 hours or more, longer than original method in the ABC-002 trial. Oral rehydration therapy is a therapy that performs prevention or treatment of dehydration by the ingestion of oral rehydration solution, which is adjusted the concentration of the electrolyte and glucose to absorb good efficiency from the gastrointestinal tract. Oral rehydration therapy (ORT) is a therapy that performs prevention or treatment of dehydration by the ingestion of oral rehydration solution, which is adjusted the concentration of the electrolyte and glucose to absorb good efficiency from the gastrointestinal tract. Many reports suggest ORT may substitute for infusion therapy. Herein, the investigators planned the study to examine the safety of replacing the fluid infusion by oral rehydration expecting to shorten the time to drip.

ELIGIBILITY:
Inclusion Criteria: 1. Patients with histological or cytological diagnosis of biliary tract cancer who haven't received cisplatin previously 2. Patients who is planned to receive chemotherapy including gemcitabine and cisplatin for biliary cancer for more than 12 weeks 3. Older than 20 years old 4. Eastern Cooperative Oncology Group Performance status of 0 or 1 5. Adequate main organ function 6. Fully oral intake ability to drink 500ml of solution before chemotherapy 7. Estimated life expectancy no less than 3 months 8. Written informed consent

- Exclusion Criteria: 1. Patients who received cisplatin previously 2. Radiological and clinical evidence of pulmonary fibrosis or interstitial pneumonia 3. Patients with uncontrolled diabetes mellitus or severe liver dysfunction or unstable angina or myocardial infarction within 3 months 4. Patients with serious infection 5. Pregnant or lactating female or patients who wish pregnant 6. Patients having severe allergy 7. Patients with other serious comorbid diseases 8. Patients with severe psychological disease 9. Patients with uncontrollable watery diarrhea 10. Patients with moderate or severe ascites /pleural effusion 11. Patients with severe psychological disease 12. Patients who are positive for a test of hepatitis B virus surface antigen (HBs antigen) without controlled with entecavir 13. Patients who is judged as an inappropriate case by the investigator

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05-22 (Actual); Primary Completion 2016-01-07 (Actual); Study Completion 2016-07-07 (Actual)

PRIMARY OUTCOMES:
Completion rate during the 12 weeks in the short hydration group | 12 weeks
  Completion rate during the 12 weeks in the short hydration group is defined as percentage proportion of treatment complete cases for 12 weeks of the eligible cases. Treatment completion is defined as carrying out a short hydration regimen via ORT.

SECONDARY OUTCOMES:
Rate of renal toxicity | 12 weeks
Adverse events | 12 weeks
Marker of renal function | 12 weeks
Response rate | 12 weeks
Time to treatment failure | 6 months
Progression free survival | 6 months
Overall survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Nagano, MD, PhD, Study Director — Osaka University Graduate School of Medicine
Locations (1):
- Osaka University, Graduate School of Medicine, Osaka, Japan